CLINICAL TRIAL: NCT02154763
Title: A Pilot Study to Assess the Feasibility of a Future Randomized, Double-Blinded, Placebo-Controlled Trial to Investigate the Role of Intra-Peritoneal Ropivacaine in Gastric Bypass Surgery: INOPAIN Trial
Brief Title: The Use of Intraperitoneal Ropivacaine in Bariatric Bypass Surgery
Acronym: INOPAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 717602410
Record Dates: First submitted 2014-05-16; First posted 2014-06-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; Bariatrics; Local anesthetic; Ropivacaine; Intraperitoneal
MeSH Terms: interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraperitoneal Normal Saline (Placebo Comparator): Intraperitoneal Normal Saline: 100mL (Milliliter) normal saline administered as in intervention arm
  Interventions: Drug: Normal Saline
- Intraperitoneal ropivacaine (Experimental): The abdomen will be entered and trocars placed in the usual manner. Using a standard suction/irrigation device and tubing, 200mg of Ropivacaine (0.2% Ropivacaine in 100mL Normal Saline) will be instilled into the abdomen at the start of the case, prior to dissection as follows. Under direct visualization, 50mL (Milliliter) (of the 100mL) will be infused over the esophageal hiatus. The remaining 50mL will be infused throughout the abdomen. The infusion line will then be flushed with 30mL (Milliliter) of Normal Saline to ensure the entire treatment dose is delivered, and no Ropivacaine remains in the tubing. The remainder of the surgery will proceed as usual.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: NAROPIN®; 84057-95-4
  Arms: Intraperitoneal ropivacaine
Drug: Normal Saline
  Other Names: Sodium Chloride; 7647-14-5
  Arms: Intraperitoneal Normal Saline

SUMMARY:
This is a pilot study in a randomized, controlled, double-blinded format and will evaluate the ability of a local anesthetic, Ropivacaine, to decrease pain after gastric bypass surgery. The drug will be administered into the abdomen during a bariatric bypass surgery. After surgery, patients who received Ropivacaine will be compared to those without Ropivacaine to determine its effect on reducing pain, recovery of lung function, ability to walk, and quality of life during recovery.

DETAILED DESCRIPTION:
Introduction: Postoperative pain control remains a major challenge for surgical procedures, including laparoscopic gastric bypass. Pain management is particularly relevant in obese patients who experience a higher number of of cardiovascular and pulmonary events. effective pain management may reduce their risk of serious postoperative complications, such as deep venous thrombosis and pulmonary emboli. The objective of this study is to evaluate the efficacy of intraperitoneal local anaesthetic, ropivacaine, to reduce postoperative pain in patients undergoing laparoscopic Roux-en-Y gastric bypass.

Methods and Analysis: A randomized controlled trial will be conducted to compare intraperitoneal ropivacaine (Intervention) versus normal saline (placebo) in 120 adult patients undergoing bariatric surgery. Ropivacaine will be infused over the oesophageal hiatus and throughout the abdomen. Patients in the control arm will undergo the same treatment as normal saline. The primary end point will be postoperative pain at 1, 2 and 4 hours postoperatively. Pain measurements will then occur every 4 hours for 24 h and every 8h until discharge. Secondary endpoints will include opioid use, peak expiratory flow, 6 min walk distance and quality of life. Intention-to-treat analysis will be used and repeated measures will be analysed using mixed model approach. post-hoc pairwise comparison of the treatment groups at different time points will be carried out using multiple comparisons with adjustments to the type 1 error. Results of the study will inform the feasibility of effectiveness of intraperitoneal ropivacaine.

Ethics and dissemination This study has been approved by the Ottawa Health Science Network Research Ethics Board and Health Canada in April 2014. The findings of the study will be disseminated through national and international conferences and peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Roux-en-Y gastric bypass surgery;
* Patients who able to tolerate general anesthetic and pneumoperitoneum;
* Patients who able to provide informed consent for the surgery;
* Patients over the age of 18 years;

Exclusion Criteria:

* Patient undergoing planned Sleeve Gastrectomy (inta-op conversion to Sleeve Gastrectomy after delivery of intraperitoneal ropivacaine will be included and analyzed using intention-to-treat approach)
* Patients with an allergy to local anesthetics
* Patients with severe underlying cardiovascular disease (ie: congestive heart failure, conduction abnormalities, and ischemic heart disease)
* Patients with chronic renal disease Stage 3 or greater (Creatinine clearance less than 60mL/hr (millilitre per hour))
* Patients with hepatic dysfunction Child-Pugh Class B or C
* Patients with previous foregut surgery including esophageal, gastric, liver, and pancreas resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mamazza, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jarrar A, Eipe N, Wu R, Neville A, Yelle JD, Mamazza J. Effect of intraperitoneal local anesthesia on enhanced recovery outcomes after bariatric surgery: a randomized controlled pilot study. Can J Surg. 2021 Nov 10;64(6):E603-E608. doi: 10.1503/cjs.017719. Print 2021 Nov-Dec. PMID 34759045
- [Derived] Wu R, Haggar F, Porte N, Eipe N, Raiche I, Neville A, Yelle JD, Ramsay T, Mamazza J. Assessing the feasibility of a randomised, double-blinded, placebo-controlled trial to investigate the role of intraperitoneal ropivacaine in gastric bypass surgery: a protocol. BMJ Open. 2014 Aug 11;4(8):e005823. doi: 10.1136/bmjopen-2014-005823. PMID 25113556

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraperitoneal Normal Saline: Intraperitoneal Normal Saline: 100mL normal saline administered as in intervention arm prior to dissection.
- Intraperitoneal Ropivacaine: 200mg of Ropivacaine (0.2% Ropivacaine in 100mL Normal Saline) prior to dissection.
Period: Overall Study
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Started | 60 | 60
Completed | 46 | 46
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (9.44) | 44.4 (9.42) | 44.75 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: Participants]
  Canada | 46 | 46 | 92
Mean BMI [Mean (Standard Deviation); unit: kg/m^2] | 45.82 (6.57) | 48.57 (6.07) | 47.195 (6.32)
History of Pain Syndromes [Number; unit: Participants] — Information collected Preoperatively and data indicates the number of participants who had Pain syndromes.
  Participants | 9 | 2 | 11
History of Asthma [Number; unit: Participants] | 6 | 14 | 20
History of Cardiovascular Disease [Number; unit: participants] | 24 | 15 | 39
History of Arthritis [Number; unit: participants] | 22 | 22 | 44
On Diabetic Medications [Number; unit: participants] | 18 | 12 | 30
On Pain Medications [Number; unit: participants] | 22 | 20 | 42
Previous Caesarean section [Number; unit: participants] | 12 | 9 | 21
Previous Laparoscopic Cholecystectomy [Number; unit: participants] | 9 | 13 | 22
Prior Surgery [Number; unit: participants] | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: 0-1 h Postoperative Pain Level
Description: Measured by the Numeric Pain Rating Scale (NRS) with a range of 0-10 where 0 represents No pain at all ( best outcome) and 10 represents Worst possible pain (worst outcome).
Time Frame: 0-1 hours post operatively
Population: Overall Number of Participants Analyzed is not consistent with numbers provided Participant Flow module due to patients refusing or being unable to provide the reading for outcome during the allocated time frame which could vary the number of results obtained in a specific time frame.
  The analysis was done and revised by our Statistician
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 42 | 45
units on a scale | 3.9762 (2.5191) | 4.3149 (2.1074)

2. Primary Outcome: 1-2 h Postoperative Pain Level
Description: as for outcome 1
Time Frame: 1-2 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 41 | 45
units on a scale | 3.5307 (1.6086) | 3.6911 (1.522)

3. Primary Outcome: 2-4 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 2-4 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intraperitoneal Normal Saline: Intraperitoneal Normal Saline: 100mL normal saline administered as in intervention arm
  Normal Saline
- Intraperitoneal Ropivacaine: The abdomen will be entered and trocars placed in the usual manner. Using a standard suction/irrigation device and tubing, 200mg of Ropivacaine (0.2% Ropivacaine in 100mL Normal Saline) will be instilled into the abdomen at the start of the case, prior to dissection as follows. Under direct visualization, 50mL (of the 100mL) will be infused over the esophageal hiatus. The remaining 50mL will be infused throughout the abdomen. The infusion line will then be flushed with 30mL of Normal Saline to ensure the entire treatment dose is delivered, and no Ropivacaine remains in the tubing. The remainder of the surgery will proceed as usual.
  Ropivacaine
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 43 | 46
units on a scale | 3.2733 (1.3186) | 3.1978 (1.1836)

4. Primary Outcome: 4-8 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 4-8 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 43 | 45
units on a scale | 3.6507 (1.7729) | 3.8387 (1.6156)

5. Primary Outcome: 8-12 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 8-12 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 45
units on a scale | 3.7955 (2.0667) | 3.9056 (1.6866)

6. Primary Outcome: 12-16 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 12-16 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 43 | 45
units on a scale | 3.4419 (2.2152) | 3.9444 (1.9283)

7. Primary Outcome: 16-20 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 16-20 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 46 | 46
units on a scale | 3.4186 (1.899) | 3.8081 (1.6071)

8. Primary Outcome: 20-24 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 20-24 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 43
units on a scale | 3.2386 (1.6548) | 3.4651 (1.5976)

9. Primary Outcome: 24-32 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 24-32 hours post operatively
Population: Overall Number of Participants Analyzed is not consistent with numbers provided Participant Flow module due to patients being discharged from hospital early or refusing reading; varying the number of results obtained in a specific time frame.
  The analysis was done and revised by our Statistician
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 37 | 38
units on a scale | 3.2568 (1.7858) | 3.1974 (1.9951)

10. Primary Outcome: 32-40 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 32-40 hours post operatively
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 35 | 38
units on a scale | 2.8143 (1.7409) | 2.9955 (1.9079)

11. Primary Outcome: 40-48 Hours Post Operative Pain Level
Description: as for outcome 1
Time Frame: 40-48 hours post operatively
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 31 | 33
units on a scale | 2.7661 (1.9842) | 2.9394 (1.3507)

12. Secondary Outcome: 1h Peak Expiratory Flow (PEF) Score
Description: Measured using the Mini Wright Peak flow meter with a range of 60-800 L/Min where 60 L/Min represents the worst possible score and 800 L/Min represents the best possible score. Value recorded is based on an average of 3 readings at every time point.
Time Frame: 1 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 42 | 45
L/min | 202.9 (99.9948) | 200.3 (88.4809)

13. Secondary Outcome: 2h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 2 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 42 | 45
L/min | 243 (104.1) | 239.8 (84.9128)

14. Secondary Outcome: 4h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 4 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 43 | 46
L/min | 251.9 (93.5798) | 256.1 (77.5092)

15. Secondary Outcome: 8h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 8 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 43 | 45
L/min | 250.9 (81.9403) | 255.3 (86.4081)

16. Secondary Outcome: 12h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 12 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 45
L/min | 240 (88.7052) | 241.6 (73.7843)

17. Secondary Outcome: 16h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 16 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 46
L/min | 233.4 (86.6212) | 242.2 (76.4464)

18. Secondary Outcome: 20h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 20 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 43
L/min | 246 (97.9415) | 245.1 (66.3817)

19. Secondary Outcome: 24h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 24 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 44 | 43
L/min | 255.2 (92.1195) | 253.8 (73.1017)

20. Secondary Outcome: 32h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 32 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 37 | 37
L/min | 256.62 (95.183) | 265.5 (84.941)

21. Secondary Outcome: 40h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 40 hours post operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 35 | 37
L/min | 255.3 (96.6315) | 265.8 (81.654)

22. Secondary Outcome: 48h Peak Expiratory Flow (PEF) Score
Description: as for outcome 12
Time Frame: 48 hours post operatively
Population: Overall Number of Participants Analyzed is not consistent with numbers provided Participant Flow module due to patients refusing, early Discharge or being unable to provide the reading for outcome during the allocated time frame which could vary the number of results obtained in a specific time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 16 | 19
L/min | 285.3 (97.1162) | 285.3 (84.6803)

23. Secondary Outcome: 6 Minute Walking Distance Post Operative Day 1 (POD1)
Description: 6-Minute walk distance (6MWD)-Defined as the distance in (m) an individual is able to walk a long a flat 30 m walkway over six--minute period, with breaks as required. walk testing has been validated in the obese population, clinically significant differences occur when distances of at least 80m occur. 0 m would be the worst possible value for this outcome and the higher the number achieved in the six-minute duration the better (Better outcome)
Time Frame: Post operative day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 42 | 46
Meters | 205.8 (94.3378) | 182.4 (97.1065)

24. Secondary Outcome: 6 Minute Walking Distance Post Operative Day 2 (POD2)
Description: as for outcome 23
Time Frame: Post operative day 2
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 36 | 38
Meters | 260 (87.8853) | 217.2 (101.7)

25. Secondary Outcome: Postoperative Day 1 Quality of Recovery Questionnaire (QR-40)
Description: 40-item questionnaire provides a global score(Minimum-score 40, Maximum-Score 200, Higher score represent better Quality of recovery of participant in both global and subscores) subscores(summed to total the global score) across five dimensions explained below, in all categories minimum score is 1, maximum score of 5 for each question.unit is scores on a scale for all questions.
  Emotional_State:9 questions subscore can range between 9-45 Physical_Comfort:12 questions, subscore range between 12-60 Psychological Support:7 questions, subscore range between 7-35 Physical_Independence:5 questions, subscore range between 5-25 Pain:7 questions, subscore range between 5-25
  Questionnaire has two parts A and B, In part A, a score of 1 represents the answer of "None of the time (Poor)"and 5 represents the answer"All of the time (Excellent)"Part B, score of 1 represents the answer"All of the time (Excellent)" and 5 represents"None of the time (Poor)
Time Frame: Post operative day 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 46 | 46
Scores on a scale | 163 (16.4944) | 163.6 (14.6931)

26. Secondary Outcome: 0-1 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to the patient
Time Frame: 0-1 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 72.2222 (206.6) | 49.2391 (192.7)

27. Secondary Outcome: 0-1 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 0-1 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 5 (7.8335) | 6.413 (8.6707)

28. Secondary Outcome: 0-1 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 0-1 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 1008.9 (951.5) | 925 (641.8)

29. Secondary Outcome: 0-1 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 0-1 h Postoperative Tramadol consumption
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 3.3333 (12.6131) | 2.1739 (10.3092)

30. Secondary Outcome: 0-1 h Postoperative Fentanyl Consumption
Description: The amount in mcg of Fentanyl administered to patient
Time Frame: 0-1 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mcg | 45.5556 (43.722) | 42.9348 (45.5409)

31. Secondary Outcome: 1-2 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to patient
Time Frame: 1-2 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 144.2 (272.9) | 141.3 (271.1)

32. Secondary Outcome: 1-2 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 1-2 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 2.3333 (6.3604) | 2.3913 (5.3478)

33. Secondary Outcome: 1-2 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 1-2 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 291.1 (488.9) | 489.1 (582.8)

34. Secondary Outcome: 1-2 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 1-2 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 9.4444 (19.43) | 8.6957 (19.1612)

35. Secondary Outcome: 1-2 h Postoperative Fentanyl Consumption
Description: The amount in mcg of Fentanyl administered to patient
Time Frame: 1-2 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mcg | 10 (17.9962) | 7.6087 (16.5576)

36. Secondary Outcome: 2-4 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to patient
Time Frame: 2-4 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 216.4 (309.6) | 240.2 (317.2)

37. Secondary Outcome: 2-4 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 2-4 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 3.2222 (6.9213) | 1.0087 (3.7421)

38. Secondary Outcome: 2-4 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 2-4 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 415.6 (604.5) | 484.8 (707.4)

39. Secondary Outcome: 2-4 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 2-4 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 12.2222 (21.7307) | 15.2174 (23.2608)

40. Secondary Outcome: 2-4 h Postoperative Fentanyl Consumption
Description: The amount in mcg of Fentanyl administered to patient
Time Frame: 2-4 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mcg | 4.4444 (13.3663) | 33.1522 (191.6)

41. Secondary Outcome: 4-12 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to patient
Time Frame: 4-12 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 1140.9 (441.5) | 1187 (394.9)

42. Secondary Outcome: 4-12 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 4-12 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 6.8889 (11.2961) | 5.2174 (9.065)

43. Secondary Outcome: 4-12 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 4-12 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 81.1111 (38.86) | 85.8696 (31.0252)

44. Secondary Outcome: 4-12 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 4-12 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 2000 (1714.1) | 1830.4 (2018.1)

45. Secondary Outcome: 12-24 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to patient
Time Frame: 12-24 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 1921.1 (414.7) | 1837 (460.7)

46. Secondary Outcome: 12-24 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 12-24 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 6.3333 (11.3016) | 5.5435 (10.1778)

47. Secondary Outcome: 12-24 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 12-24 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 141.1 (38.86) | 138 (31.9458)

48. Secondary Outcome: 12-24 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 12-24 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 2066.7 (1923.5) | 2760.9 (3085.3)

49. Secondary Outcome: 24-48 h Postoperative Tylenol Consumption
Description: The amount in mg of Tylenol administered to patient
Time Frame: 24-48 hours post operatively
Population: as for outcome 22
Measure: Median (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 3033.3 (1239.5) | 2826.1 (1330.1)

50. Secondary Outcome: 24-48 h Postoperative Ketorolac Consumption
Description: The amount in mg of Ketorolac administered to patient
Time Frame: 24-48 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 2.3333 (7.8044) | 3.2609 (8.8955)

51. Secondary Outcome: 24-48 h Postoperative Tramadol Consumption
Description: The amount in mg of Tramadol administered to patient
Time Frame: 24-48 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 216.7 (97.1175) | 215.2 (101.6)

52. Secondary Outcome: 24-48 h Postoperative Dilaudid Consumption
Description: The amount in mg of Dilaudid administered to patient
Time Frame: 24-48 hours post operatively
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 45 | 46
mg | 2933.3 (3563.7) | 3000 (3489.7)

53. Secondary Outcome: Postoperative Day 7-10 Quality of Recovery Questionnaire (QR-40)
Description: 40-item questionnaire provides a global score(Minimum-score 40,Maximum-Score 200, Higher score represent better Quality of recovery of participant in both global and subscores) subscores(summed to total the global score) across five dimensions explained below, in all categories minimum score is 1,maximum score of 5 for each question.unit is scores on a scale for all questions.
  Emotional_State:9 questions subscore can range between 9-45 Physical_Comfort:12 questions, subscore range between 12-60 Psychological Support:7 questions, subscore range between 7-35 Physical_Independence:5 questions, subscore range between 5-25 Pain:7 questions,subscore range between 5-25
  Questionnaire has two parts A and B, In part A, a score of 1 represents the answer of "None of the time (Poor)"and 5 represents the answer"All of the time (Excellent)"Part B, score of 1 represents the answer"All of the time (Excellent)" and 5 represents"None of the time (Poor)
Time Frame: Post operative day 7-10
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 41 | 42
Scores on a scale | 183.5 (14.1829) | 182.7 (14.0707)

54. Secondary Outcome: 6 Minute Walking Distance Post Operative Day 7-10 (POD 7-10)
Description: as for outcome 23
Time Frame: Post operative day 7-10 (Follow-up Clinic)
Population: Overall Number of Participants Analyzed is not consistent with numbers provided Participant Flow module due to patients refusing, Missing Appointment or being unable to provide the reading for outcome during the allocated time frame which could vary the number of results obtained in a specific time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intraperitoneal Normal Saline | Intraperitoneal Ropivacaine
Number analyzed (Participants) | 41 | 44
meters | 373.3 (68.1203) | 352.4 (90.2276)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to postoperative day 7
Description: Safety end points are:
  * Serious adverse event (SAE) rates
  * Surgical complication rates
  Anticipated SAEs include the risks of an anaesthetic, bleeding, wound infection, bowel injury, unexpected leak, pneumothorax, obstruction and general complications such as a thromboembolic events, pneumonia, cardiac events and stroke.
  Adverse events are collected on regular intervals until postoperative day 7
Groups:
- Control: Intraperitoneal Saline: 100mL normal saline administered as in intervention arm
Arm/Group | Control | Intraperitoneal Ropivacaine
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No